CLINICAL TRIAL: NCT00868023
Title: A Phase II, Multinational, Multicentre, Double Blind, Double Dummy, Randomised, 5-way Cross-over, Placebo and Active Controlled Clinical Study to Test the Non-inferiority of a Single Dose of CHF 1535 (Fixed Combination of Beclomethasone Dipropionate 100 µg Plus Formoterol Fumarate 6 µg Dry Powder) Via NEXT™ DPI 1 or 4 Inhalations Versus CHF 1535 (Beclomethasone Dipropionate 100 µg Plus Formoterol Fumarate 6 µg) pMDI With HFA-134a Propellant 1 or 4 Puffs on FEV1 AUC0-12h in Partly Controlled Adult Asthmatic Patients
Brief Title: Next DPI LABA, Multicentre, 5-way Cross-over, Adult Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Pr SD Singh, Medecines Evaluation Unit - Southmoor Road - M23 9QZ Manchester - United Kingdom
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-0809-PR-0038; 2008-004842-10 (EudraCT Number)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): CHF 1535 DPI : BDP/Formo 400/24 µg
  Interventions: Drug: CHF 1535 Next DPI
- 2 (Active Comparator): CHF 1535 pMDI HFA : BDP/Formo 400/24 µg
  Interventions: Drug: Foster BDP/Formoterol
- 3 (Experimental): CHF 1535 DPI : BDP/Formo 100/6 µg
  Interventions: Drug: CHF 1535 Next DPI
- 4 (Active Comparator): CHF 1535 pMDI HFA : BDP/Formo 100/6 µg
  Interventions: Drug: Foster BDP/Formoterol
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CHF 1535 Next DPI — CHF 1535 DPI : BDP/Formoterol : 100/6 µg (daily dose : BDP/Formoterol : 400/24 µg)
  Arms: 1
Drug: Foster BDP/Formoterol — BDP/Formoterol 100/6 µg (daily dose : BDP/Formoterol : 400/24 µg)
  Arms: 2
Drug: CHF 1535 Next DPI — CHF 1535 DPI : BDP/Formoterol : 100/6 µg (daily dose : BDP/Formoterol : 100/6 µg)
  Arms: 3
Drug: Foster BDP/Formoterol — BDP/Formoterol 100/6 µg (daily dose : BDP/Formoterol : 100/6 µg
  Arms: 4
Drug: Placebo — Placebo
  Arms: 5

SUMMARY:
Multinational, multicentre, randomised, double blind, double dummy, placebo and active controlled, 5-way cross over

DETAILED DESCRIPTION:
To demonstrate the non-inferiority in terms of FEV1 AUC0-12h between a single dose of CHF 1535 via NEXT DPI and CHF 1535 via HFA-134a "extrafine" pMDI in partly controlled adult asthmatic patients

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent obtained prior to any study-related procedures.
* Outpatient male or female aged ≥ 18 years.
* Evidence for "partly controlled" asthma in the 2 weeks before the screening visit
* Under previous inhaled corticosteroids (ICS) treatment at the screening visit
* Forced expiratory volume in the first second (FEV1) ≥ 60% and ≤ 90% of the predicted normal values at the screening visit.
* A documented positive response to the reversibility test at the screening visit, defined as ΔFEV1 ≥ 12% and ≥ 200 mL over baseline, 30 minutes after 400 μg salbutamol pMDI
* Patients free of long-acting beta2-agonists (LABAs) treatment for at least 2 weeks before the screening visit.
* Patients free of short-acting beta2-agonists (SABAs) treatment for at least 6 hours before the screening visit.
* Non-smokers or ex-smokers

Exclusion Criteria:

* Pregnant or lactating women or all women physiologically capable of becoming pregnant UNLESS they are menopausal or are using effective and acceptable methods of contraception.
* Significant seasonal variation in asthma or asthma occurring only during episodic exposure to an allergen or a chemical sensitizer.
* History of near fatal asthma (e.g. brittle asthma, hospitalisation for asthma exacerbation in Intensive Care Unit) within 1 year before screening.
* Occurrence of asthma exacerbations or respiratory tract infections in the 4 weeks preceding the screening visit.
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency.
* Diagnosis of restrictive lung disease.
* Patients treated with oral or parenteral corticosteroids in the previous 8 weeks (12 weeks for parenteral depot corticosteroids) before screening visit.
* Intolerance or contra-indication to treatment with beta2-agonists and/or inhaled corticosteroids.
* Allergy, sensitivity or intolerance to study drugs or excipients.
* Significant medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-12h | Every week

SECONDARY OUTCOMES:
FVC as assessed at the same time points as for FEV1; Peak FEV1 in terms of absolute values and % of change from baseline Safety evaluation | Every week

CONTACTS AND LOCATIONS:
Overall Officials: David Singh, Professor, Principal Investigator — Medecines Evaluation Unit - Southmoor Road - M23 9QZ Manchester - UK
Locations (1):
- Pr DS SINGH, Manchester, United Kingdom

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2008-004842-10